CLINICAL TRIAL: NCT06304259
Title: The Effect of Different Modalities of Cryotherapy on Post-Operative Pain Level in Patients With Symptomatic Irreversible Pulpitis (Randomized Control Trial)
Brief Title: Effect of Different Modalities of Cryotherapy on Post-Operative Pain in Patients With Symptomatic Irreversible Pulpitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Yara Adel Mohamed Taha, Dr, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24428
Record Dates: First submitted 2024-02-05; First posted 2024-03-12 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Endodontic Disease; Endodontically Treated Teeth
MeSH Terms: conditions — Dental Pulp Diseases; Tooth, Nonvital | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): participants will receive standard root canal treatment with final flush of normal saline at the room temperature after cleaning and shaping and before obturation.
  Interventions: Drug: Saline
- Submucosal cryotherapy infiltration (Experimental): participants will receive Submucosal infiltration injection of 1 mL cryo-treated saline maintained at a temperature of 2 to 5°C before the normal local anaesthetic routine.
  Interventions: Drug: Saline
- Intracanal cryotherapy (Experimental): participants will receive root canal treatment with final flush of cold saline maintained at a temperature of 2 to 5°C
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Saline — Submucosal infiltration injection of 1 mL cryo-treated saline maintained at a temperature of 2 to 5°C before the normal local anaesthetic routine
  Arms: Control; Submucosal cryotherapy infiltration
Drug: Saline — root canal treatment with final flush of cold saline maintained at a temperature of 2 to 5°C
  Arms: Control; Intracanal cryotherapy

SUMMARY:
Problem statement: The post-operative pain after endodontic treatment. aim of study: The study is aiming to compare postoperative pain after submucosal cold saline injection (submucosal cryotherapy) (SMC) versus intra-canal cryotherapy (ICC) in mandibular single rooted premolars with symptomatic irreversible pulpitis with symptomatic apical periodontitis (SAP). The material and methods: Subjects and methods: sixty patients will be randomly divided into three groups: the SMC group, the ICC group, and the control group. The patients' postoperative pain will be recorded at 12, 24, and 48 hours postoperatively by questioning them. Quantification of substance P will be done using an ELISA test from peri-radicular fluid swab.

ELIGIBILITY:
Inclusion Criteria:

* Older than age of 18 years
* Participants willing to commit for the entire period of the trial and Both genders
* agreed to sign the written consent after full explanation of the study
* Having a mandibular single rooted premolar tooth with vital pulp
* These patients were also suffering from symptoms of symptomatic irreversible pulpitis and apical periodontitis, intermittent or continuous sharp pain that lasts longer after removal of the stimulus. on the basis of the clinical symptoms of severe preoperative pain (visual analogue scale)

Exclusion Criteria:

* Vulnerable group; prisoners, pregnant females, mentally ill, etc…
* Teeth with open apices
* A previous root canal treatment
* Sinus tracts
* Presence of periodontal pockets >3 mm in the affected tooth

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
postoperative pain | After 12 hours
  measure intensity of post operative pain using visual analogue scale that was represented by a 100 mm horizontal ruler with no number markings other than a 0 at one end and a 10 at the other end. The following categories of postoperative pain levels were used to assess pain: 0 indicating no pain, mild pain (1-3), moderate pain (4-7) and severe pain (8-10)
postoperative pain | After 24 hours
  measure intensity of post operative pain using visual analogue scale that was represented by a 100 mm horizontal ruler with no number markings other than a 0 at one end and a 10 at the other end. The following categories of postoperative pain levels were used to assess pain: 0 indicating no pain, mild pain (1-3), moderate pain (4-7) and severe pain (8-10)
postoperative pain | After 48 hours
  measure intensity of post operative pain using visual analogue scale that was represented by a 100 mm horizontal ruler with no number markings other than a 0 at one end and a 10 at the other end. The following categories of postoperative pain levels were used to assess pain: 0 indicating no pain, mild pain (1-3), moderate pain (4-7) and severe pain (8-10)

SECONDARY OUTCOMES:
Substance P level | After 15 minutes from access cavity preparation
  Quantification of substance P will be done using an ELISA test from peri-radicular fluid swab.
Substance P level | After 30 minutes from access cavity preparation
  Quantification of substance P will be done using an ELISA test from peri-radicular fluid swab.
Substance P level | after 24 hour
  Quantification of substance P will be done using an ELISA test from peri-radicular fluid swab.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Ain shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No